CLINICAL TRIAL: NCT03299660
Title: Phase II Trial PD-L1/PD-1 Blockade Avelumab (MSB0010718C) With Chemoradiotherapy for Locally Advanced Resectable Rectal Cancer
Brief Title: Avelumab With Chemoradiation in Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AveRec
Record Dates: First submitted 2017-09-24; First posted 2017-10-03 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — avelumab; Fluorouracil; Capecitabine; Radiotherapy

STUDY DESIGN:
Intervention Model Description: All participants will receive standard LCCRT treatment followed by 4 cycles of Avelumab followed by surgical resection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): Long course chemoradiotherapy (LCCRT) comprised of 50.4 Gy radiotherapy in conjunction with 5FU (225mg/m2/day continuous infusion)/Capecitabine (825 mg/m2 BID on RT days) over 5. 5 weeks, followed by 4 cycles of Avelumab. This is then followed up with surgical resection
  Interventions: Drug: Avelumab; Drug: 5 Fluorouracil; Drug: Capecitabine Pill; Radiation: Radiotherapy; Procedure: Surgical Resection

INTERVENTIONS:
Drug: Avelumab — Avelumab 10 mg/Kg every 2 weeks for 4 cycles post LCCRT
  Other Names: MSB0010718C
Drug: 5 Fluorouracil — 5FU continuous infusion 225mg/m2/day during radiotherapy
Drug: Capecitabine Pill — Can be administered in place of 5FU infusion. Dose = 825 mg/m2 twice a day on each day of radiotherapy
Radiation: Radiotherapy — 50.4 Gy in 28 fractions delivered over 5.5 weeks as 5 fractions/week
Procedure: Surgical Resection — Surgical resection of tumour mass post radiotherapy and chemotherapy

SUMMARY:
This trial is investigating the inclusion of avelumab post long-course chemo-radiotherapy in patients with resectable locally advanced rectal cancer. It is hypothesised that this may enhance the pathological and imaging response rates whilst potentially reducing the relapse rates. Participants will receive standard long course chemoradiotherapy (LCCRT) treatment with radiotherapy and 5-fluorouracil (5 FU)/Capecitabine for 6 weeks, this then followed by 4 cycles of Avelumab and then surgical resection. The trial will measure disease response just prior to surgery and participants will be followed up for a minimum of 18 months (from study entry) and up to 42 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years at screening
2. Patients with histologically confirmed rectal adenocarcinoma clinical stage T3bN1-N2M0, T3c/dN0-N2M0, T4N0-N2M0 (see Appendix 1),1 as defined by pelvic MRI
3. Planned to receive neoadjuvant long course chemoradiotherapy (50.4 Gy, with infusional 5FU or capecitabine) followed by curative total mesorectal excision plus abdomino-perineal resection or anterior resection
4. Lower border of tumour must be within 12 cm from anal verge
5. Measurable disease by RECIST1.12
6. ECOG Performance Status 0-1
7. Patients must be willing to provide fresh (where possible) and archival tumour tissue samples for translational studies at specified time points
8. Adequate organ function

   1. Absolute neutrophil count ≥1.5 x 109/L
   2. Platelet count ≥100 x 109/L
   3. Haemoglobin ≥ 90 g/L (may have been transfused)
   4. Creatinine ≤ 1.5 x upper normal limit OR measured creatinine clearance ≥ 50 mL/minute
   5. Total bilirubin ≤ 1.5 x upper normal limit
   6. AST/ALT ≤ 2.5 x upper normal limit
9. Female patients of childbearing potential must have a negative urine or serum pregnancy test at screening
10. Both male and female patients should be willing to use highly effective contraception (that is, methods with a failure rate of less than 1% per year) if the risk of conception exists
11. Has provided written informed consent for the trial
12. Agrees to comply with trial therapy or trial-related investigations and evaluations

Exclusion Criteria:

1. Patients with disease outside the pelvis
2. Prior pelvic radiotherapy
3. Participation in another interventional clinical trial within 30 days of registration (participation in observational studies are permitted)
4. Concurrent anti-cancer treatment
5. Concurrent treatment with a non-permitted drug (Section 8.3.2)
6. Major surgery for any reason within 4 weeks of registration (except defunctioning stoma creation with the patient having fully recovered from this procedure)
7. Current use of immunosuppressive medication. Except for the following: (a) intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); (b). Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; (c). Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication); (d) Short-term administration of systemic steroids (that is, for allergic reactions or the management of irAEs) is allowed while on study.

   Note: Patients receiving bisphosphonate or denosumab are eligible
8. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible
9. Active or history of immunodeficiencies
10. Has received prior therapy with an anti-PD1, anti-PDL1, anti-PDL2 or anti-CTLA-4 agents
11. Has clinically significant (that is, active) cardiovascular disease: cerebral vascular accident / stroke (< 6 months prior to registration), myocardial infarction (< 6 months prior to registration), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious cardiac arrhythmia requiring medication.
12. Has an active infection requiring systemic therapy
13. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
14. Prior malignancies within 3 years of registration (with the exception of non- melanomatous skin cancer)
15. Prior organ transplantation, including allogeneic stem-cell transplantation
16. A known history of testing positive for HIV or known acquired immunodeficiency syndrome (AIDS)
17. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test is positive)
18. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (CTCAE v4.03 grade ≥ 3)
19. Is pregnant or lactating
20. Vaccination within 4 weeks of registration and while on trials is prohibited except for administration of inactivated vaccines
21. Known deficiency of dihydropyrimidine dehydrogenase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Pathological Response rate | At time of resection i.e.16 -18 weeks post commencement of treatment
  To investigate the role of PD-L1 blockade for rectal cancer following neoadjuvant LCCRT, prior to definitive surgical resection, in terms pathological response rates. Assessed by tumour regression grade in resected rectal cancers post LCCRT at the time of definitive surgery: according to Ryan et al

SECONDARY OUTCOMES:
Response as per structural imaging | At 8 weeks post LCCRT
  Describe radiological response rate based on Pelvic MRI post PD-L1 blockade as per RECIST 1.1
Overall FDG PET response | At 8 weeks post LCCRT
  Describe FDG-PET response rate post PDL1 blockade as per PERCIST
Define toxicity during administration of PDL1 inhibitor and post-surgery | From consent until 4 weeks post surgery
  Worst grade AE's and SAE's CTCAE version 4.03
Determine rate of downstaging | At time of surgical resection
  Patients will be considered downstaged if the pathologic T or N stage at surgery assessment is lower than the initial radiological stage.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Michael, A/Prof, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (7):
- Australia (7):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore, St Leonards, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Monash Health, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria

IPD SHARING:
Plan to Share IPD: No